CLINICAL TRIAL: NCT03755505
Title: The Microbiome of Sputum, Urine and Feces in Healthy Persons and Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Clinical Professor, Asan Medical Center
Other Study IDs: 2018-0980
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema or COPD; Microbiota
Keywords: Emphysema; Microbiome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Defecation; Urination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Smoker: Healthy smoker with normal spirometry value
  Interventions: Diagnostic Test: obtain samples from sputum, feces and urine
- COPD: Patients with smoking history at least 10 pack-year Patients with persistent airflow limitation that was not fully reversible (e.g. post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) <0.7)
  Interventions: Diagnostic Test: obtain samples from sputum, feces and urine

INTERVENTIONS:
Diagnostic Test: obtain samples from sputum, feces and urine — Samples are obtained from participants. No further intervention is required. Obtained samples will be further analyzed.

SUMMARY:
Extensive studies suggest composition of microbiome of respiratory samples or lung tissues in COPD patients is different from the composition of healthy smokers. Aim of this study is to analyze composition of microbiome of various samples (e.g. feces, sputum, and urine) and to describe difference of composition between COPD patients and healthy smokers.

DETAILED DESCRIPTION:
After the introduction of the Gut-Lung axis theory, extensive studies revealed diversity of microbiomes among healthy smokers and COPD patients form the respiratory samples or lung tissues. In the previous study, distinct difference in composition of microbiome in lung tissue between healthy smokers and COPD patients was reported. This is a cross sectional study to analyze composition of microbiome of various samples (e.g. feces, sputum, and urine) and to compare difference of composition between COPD patients and healthy smokers. This study would help establishing gut-lung axis model in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with smoking history at least 10 pack-year
* Patients with persistent airflow limitation that was not fully reversible (e.g. post-bronchodilator forced expiratory volume in 1 second/forced vital capacity ( FEV1/FVC) <0.7)

Exclusion Criteria:

* Patients with co-existing illness that would interfere with study results (e.g., malignancy, congestive heart failure, cerebrovascular disorders, chronic renal failure, diabetes with severe complications, or uncontrolled hypertension)
* Patients with respiratory disease other than obstructive lung disease (e.g., previous pulmonary resection, tuberculosis-destroyed lung, and bronchiectasis)
* Patients with recent (8 weeks prior to screening) exacerbation or other respiratory illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: COPD group
  - Same as above
  Healthy smokers
  * Participants with smoking history
  * Participants with normal spirometry results
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity measured by operational taxonomic unit (OTU) quantitative analysis | An average of 1 month
  DNA is extracted from each sample from each patient by using a DNA Isolation Kit. The 16S universal primers are used for amplification of 16S ribosomal ribonucleic acid (rRNA) genes with polymerase chain reaction (PCR) system. After amplication, sequencing is performed using the GREENGENES database, after which a metagenomic analysis was performed by the MD Healthcare corporation using MDx-Pro software (Ver.1, Seoul, South Korea). Taxonomic assignment of these sequences is carried out with an operational taxonomic unit (OTU) cutoff of 3%.
Microbiome composition by metagenomic analysis | An average of 1 month
  The composition of microbiome is presented as bar graph.

SECONDARY OUTCOMES:
Biodiversity described by the Shannon diversity index and the Simpson index | An average of 1 month
  The Shannon index and the Simpson index is calculated by using metagenomic data.
Biodiversity described by Principal Component Analysis (PCA) | An average of 1 month
  PCA is performed for all 16S rRNA gene reads clustered at a 97% similarity.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Kim YS, Kim KH, Choi JP, Kim YK, Yun S, Sharma L, Dela Cruz CS, Lee JS, Oh YM, Lee SD, Lee SW. The microbiome of the lung and its extracellular vesicles in nonsmokers, healthy smokers and COPD patients. Exp Mol Med. 2017 Apr 14;49(4):e316. doi: 10.1038/emm.2017.7. PMID 28408748
- [Background] Marsland BJ, Trompette A, Gollwitzer ES. The Gut-Lung Axis in Respiratory Disease. Ann Am Thorac Soc. 2015 Nov;12 Suppl 2:S150-6. doi: 10.1513/AnnalsATS.201503-133AW. PMID 26595731
- [Background] Pragman AA, Kim HB, Reilly CS, Wendt C, Isaacson RE. The lung microbiome in moderate and severe chronic obstructive pulmonary disease. PLoS One. 2012;7(10):e47305. doi: 10.1371/journal.pone.0047305. Epub 2012 Oct 11. PMID 23071781
- [Background] Erb-Downward JR, Thompson DL, Han MK, Freeman CM, McCloskey L, Schmidt LA, Young VB, Toews GB, Curtis JL, Sundaram B, Martinez FJ, Huffnagle GB. Analysis of the lung microbiome in the "healthy" smoker and in COPD. PLoS One. 2011 Feb 22;6(2):e16384. doi: 10.1371/journal.pone.0016384. PMID 21364979
- [Derived] Lee SH, Kim J, Kim NH, Kim OH, Shon CH, Kim SJ, Jang Y, Yun S, Lim SE, Jung SY, Yoo HJ, Heo SH, Lee SW. Gut microbiota composition and metabolite profiling in smokers: a comparative study between emphysema and asymptomatic individuals with therapeutic implications. Thorax. 2023 Nov;78(11):1080-1089. doi: 10.1136/thorax-2021-217923. Epub 2023 Jul 26. PMID 37495367